CLINICAL TRIAL: NCT00052065
Title: Phase 1-2a Dose-Ranging Study of TLK286 in Combination With Doxil in Platinum Refractory or Resistant Ovarian Cancer
Brief Title: TLK286 in Combination With Doxil in Platinum Refractory or Resistant Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Gail Brown, M.D. Chief Medical Officer, Telik, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.2011
Record Dates: First submitted 2003-01-21; First posted 2003-01-23 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-06

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — TER 286

INTERVENTIONS:
Drug: TLK286

SUMMARY:
This is a dose-ranging, open-label, Phase 1-2a study of TLK286 in combination with Doxil in patients with platinum refractory or resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of epithelial cancer of the ovary, fallopian tube cancer or primary peritoneal cancer
* Recurrent epithelial ovarian cancer or persistent disease following primary treatment
* At least one, but no more than four, prior platinum-containing chemotherapy regimens
* At least one prior taxane-containing regimen

Exclusion Criteria

* A history of prior malignancy except for adequately treated carcinoma in situ of the uterine cervix, basal cell or squamous cell skin cancer, or other cancer for which the patient has been disease-free for 2 years
* Known leptomeningeal metastases or carcinomatous meningitis
* Have received prior Doxil or other liposomal doxorubicin
* Having received whole pelvis radiation therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2003-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kavanagh JJ, Levenback CF, Ramirez PT, Wolf JL, Moore CL, Jones MR, Meng L, Brown GL, Bast RC Jr. Phase 2 study of canfosfamide in combination with pegylated liposomal doxorubicin in platinum and paclitaxel refractory or resistant epithelial ovarian cancer. J Hematol Oncol. 2010 Mar 11;3:9. doi: 10.1186/1756-8722-3-9. PMID 20222977